CLINICAL TRIAL: NCT00417807
Title: Open-label Trial of Imatinib Mesylate in Patients With Refractory Desmoplastic Small Round Cell Tumors (DSRCT) Expressing PDGF-R
Brief Title: Imatinib Mesylate in Patients With Refractory Desmoplastic Small Round Cell Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BIT06
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Refractory Desmoplastic Small Round Cell Tumors
Keywords: refractory desmoplastic small round cell tumors; PDGF-R
MeSH Terms: interventions — Imatinib Mesylate

ARMS (1):
- Gleevec/Glivec (Experimental)
  Interventions: Drug: Imatinib mesilate

INTERVENTIONS:
Drug: Imatinib mesilate
  Other Names: STI571

SUMMARY:
An open-label, non-comparative study conducted to investigate the activity and safety of imatinib mesylate in refractory desmoplastic small round cell tumors expressing PDGF-R. Patients will be treated up to 12 months, or to disease progression. Tumor will be evaluated according to Recist criteria

ELIGIBILITY:
Inclusion criteria:

1. Patients > 16 years of age.
2. Histologically documented diagnosis of DSRCT, unresponsive or in no complete remission after any conventional multimodality approach.
3. Immunohistochemical documentation of activated PDGF-R expression by tumor
4. At least one measurable site of disease
5. Performance status 0,1, 2 or 3 (Eastern Cooperative Oncology Group)
6. Adequate end organ function

Exclusion criteria:

1. Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Patient is < 5 years free of another primary malignancy
3. Patient with congestive heart failure or myocardial infarction within 6 months of study
4. Female patients who are pregnant or breast-feeding.
5. Severe and/or uncontrolled medical disease
6. Known brain metastasis.
7. Chronic active hepatitis or cirrhosis
8. Known diagnosis of human immunodeficiency virus (HIV) infection.
9. Chemotherapy within 4 weeks prior to study entry, unless the disease is rapidly progressing.
10. Previous radiotherapy to > 25 % of the bone marrow
11. Major surgery within 2 weeks prior to study entry.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Overall tumor response rates | Assessed every 3 months
  An imaging technique (CT scan or MRI) determined tumor response according to RECIST criteria.

SECONDARY OUTCOMES:
Explore how Imatinib cooperated with other treatment modatilities | Survival data was collected until death
  Recorded survival after treatment and other associated treatment modalities.
Safety and tolerability | Safety data collected until patients were no longer in study
Conversion rate to surgical resectability | After best tumor response.
  Assessed actual resectability rate after therapy compared to resectability before therapy.
Mutational analysis of molecular targets of imatinib (at any time during the study) | At any time during the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (8):
- Italy (8):
  - Novartis Investigative Site, Ivrea
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Ravenna
  - Novartis Investigative Site, Rozzano
  - Novartis Investigative Site, Torino
  - Novartis Investigative Stie, Vatania